CLINICAL TRIAL: NCT05682586
Title: Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cells in the Treatment of Severe and Critical COVID-19 Patients
Brief Title: UC-MSCs in the Treatment of Severe and Critical COVID-19 Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFSC-2022(CR)-05
Record Dates: First submitted 2023-01-08; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Mesenchymal Stem Cell; COVID-19 Pneumonia
Keywords: covid-19 pneumonia; umbilical cord mesenchymal stem cells
MeSH Terms: interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- standard therapy (No Intervention): Participants will receive standard therapy, including oxygen therapy，glucocorticoid and other antiinflammatory drugs and supportive treatments according the ninth edition of Chinese guidelines for the treatment of COVID-19 infection.
- Paxlovid treatment (Active Comparator): Participants will receive paxlovid treatment on the basis of standard therapy.
  Interventions: Drug: paxlovid
- UC-MSCs treatment (Experimental): Participants will receive two doses of UC-MSCs instillation at the first and fourth day after the assignment.
  Interventions: Biological: umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cells — Participants will receive two doses of UC-MSCs treatment, each dose will contain 1*10^6 cells/kg suspended in 100 ml albumin solution.
  Arms: UC-MSCs treatment
Drug: paxlovid — Participants will receive standard dose of paxlovid therapy, which contains 300mg namatevir and 100mg litonavir twice a day for a total course of 5 days.
  Arms: Paxlovid treatment

SUMMARY:
The goal of this randomized, controlled, open-labeled interventional clinical trial is to test the efficacy and safety of umbilical cord mesenchymal stem cells (UC-MSCs) in the treatment of severe and critical COVID-19 patients. The main questions it aims to answer are: 1. The efficacy of UC-MSCs in the treatment of severe and critical COVID-19 patients. 2. The safety of UC-MSCs in the treatment of severe and critical COVID-19 patients. 3. The potential immune mechanisms of UC-MSCs in the treatment of severe and critical COVID-19 patients. Participants will receive standard therapy, Paxlovid treatment or the UC-MSCs treatment. For the standard treatment, it will be conducted according the 9th edition of Chinese guidelines for COVID-19 infection. For UC-MSCs treatment, participants will be given UC-MSCs instillation at the first and fourth day after assignment. Blood examples will be taken at indicated time for arterial blood gas analysis and other tests. And participants should also objectively report their symptoms change and other information related to the treatment as listed the research protocol.

ELIGIBILITY:
Inclusion Criteria:

* The age ranges from 18 to 75 (inclusive), regardless of gender.
* Patients diagnosed with severe and critical COVID-19 pneumonia within one week, according to the Chinese diagnostic criteria for COVID-19 pneumonia in the Diagnosis and Treatment Plan for COVID-19 Pneumonia (Tentative Ninth Edition).
* 20kg/m2≤body mass index（BMI）≤30 kg/m2.
* Volunteer to participate in this clinical study and sign the written informed consent.

Exclusion Criteria:

* Those who are using immunosuppressive drugs or long-term immunosuppressive drugs after organ transplantation.
* T lymphocyte abnormality (allogeneic may be considered, depending on clinical opinion), HIV positive.
* Highly allergic or have a history of severe allergy, especially Interleukin-2 allergy.
* Pregnant and lactating women.
* Patients with severe autoimmune disease history; Allergies to all biological reagents in this treatment, such as Interleukin-2.
* Patients with serious complications, including chronic cardiac insufficiency (NYHA cardiac function grading assessment of cardiac function grade III - IV), chronic renal insufficiency (CKD stage 3 and above); Chronic liver insufficiency (Child-Pugh score>7); Patients with malignant tumors.
* Patients with pulmonary embolism or acute coronary syndrome.
* Patients with severe organ dysfunction caused by other diseases.
* There are other situations that the researcher thinks are not suitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index | Change from baseline Oxygenation index (PaO2/FiO2) at 1,3,7,14,28 (or before the day of discharge if participants discharge within 28 days) days after the treatment.
  Oxygenation index is the artery partial pressure of oxygen divided by the concentration of inhaled oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: liu zhongming, Dr., Study Chair — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided